CLINICAL TRIAL: NCT05587751
Title: Evaluating the Impact of Gender-Affirming Treatments on Pulmonary Function in Transgender and Gender Diverse (TGD) Patients
Brief Title: Evaluation of Gender-Affirming Treatments on Pulmonary Function in Transgender and Gender Diverse Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gustavo A. Cortes Puentes, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-007173
Record Dates: First submitted 2022-09-27; First posted 2022-10-20 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Hormonal Gender-Affirming Therapy
MeSH Terms: interventions — Spirometry; Plethysmography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pulmonary Function in Transgender and Gender Diverse Patients (Experimental): Transgender and gender diverse (TGD) patients undergoing masculinizing or feminizing hormone therapies will have breathing tests to evaluate their lung function
  Interventions: Diagnostic Test: Spirometry; Diagnostic Test: Plethysmography

INTERVENTIONS:
Diagnostic Test: Spirometry — Pulmonary function test to measure lung function
Diagnostic Test: Plethysmography — Pulmonary function test to measure lung volume

SUMMARY:
The purpose of this research study is to evaluate whether undergoing gender affirming care will impact the way the lungs function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects speaking any language will be offered participation.
* Subjects capable of providing informed consent to the study. For those subjects younger than 18 years old who agree to participate in the study, informed consent will be obtained from patient's parents/guardian.
* Subjects capable of performing pulmonary function test (PFT) maneuvers, as per pulmonary function test laboratory protocol.
* Patients will be enrolled through the Mayo Clinic Rochester Transgender and Intersex
* Specialty Care Clinic (TISCC), once patient has decided to undergo hormonal gender-affirming therapies (pubertal blockers, and masculinizing or feminizing hormone therapies).

Exclusion Criteria:

* Subjects unable to provide consent, or subjects who do not agree to discuss the study with their parents/guardians.
* The presence of contraindications for pulmonary function testing including (these will be reviewed at the time of recruitment and prior to each spirometry associated with the study):

  * Recent surgical procedures (<3 months) that could be affected by lung function testing, including the following categories: Abdominal surgery, Eye surgery, Thoracic surgery, Ear surgery, Brain surgery, Vascular surgery.
  * The presence of previously known respiratory disorders including pulmonary embolism (<6 months), pleural effusion, pneumothorax, hemoptysis.
  * Recent myocardial infarction (<1 month), new cardiac arrythmia (<3 months), recent cardiac pacemaker implantation (<3 months).
  * Heart failure symptoms, significant shortness of breath, tachycardia, or angina
* The presence of chronic pulmonary diseases that maybe associated with changes in pulmonary function overtime such as asthma, chronic obstructive pulmonary disease, or interstitial lung diseases.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in lung volume (Total Lung Capacity, Vital Capacity, Functional Residual Capacity, Residual Volume) | Baseline, 6-month Follow-Up, 12-month Follow-Up, 18-month Follow-Up
  The longitudinal changes in lung volumes after both masculinizing and feminizing hormone therapy in transgender and gender diverse (TGD) patients.
Change in forced expiratory volume | Baseline, 6-month Follow-Up, 12-month Follow-Up, 18-month Follow-Up
  Measured by spirometry to determine the volume of air that can be exhaled in 1 second with a forced breath
Change in forced vital capacity | Baseline, 6-month Follow-Up, 12-month Follow-Up, 18-month Follow-Up
  Measured by spirometry to determine the maximal amount of air that can be forcibly exhaled from the lungs after a full inhale, reported as liters (L)
Change in peak expiratory flow | Baseline, 6-month Follow-Up, 12-month Follow-Up, 18-month Follow-Up
  Measured by a peak flow meter is the maximum forced expiratory flow, reported in liter per minute (L/min)
Change in maximal mid-expiratory flow rate | Baseline, 6-month Follow-Up, 12-month Follow-Up, 18-month Follow-Up
  Measured by spirometry to determine the rate of airflow where half of the forced vital capacity is exhaled

SECONDARY OUTCOMES:
Time of "gender adjustment" of PFT's normative values | Baseline, 6-month Follow-Up, 12-month Follow-Up, 18-month Follow-Up
  The time of "gender adjustment" of PFT's normative values (PFTs results correlate most closely with patient's gender than with their sex-assigned at birth) in response to gender-affirming hormone therapy in transgender and gender diverse (TGD) patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Cortes Puentes, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No